CLINICAL TRIAL: NCT02073630
Title: Contribution du Cervelet Dans l'Adaptation Sensori-motrice Via Les Oscillations Gamma : le Cas de la Dystonie
Brief Title: Contribution of the Cerebellum In Sensory-motor Adaptation Via Gamma Oscillations: the Case of Dystonia
Acronym: GAMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C13-45
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-08

CONDITIONS: Primary Dystonia
Keywords: magnetoencephalography; non invasive brain stimulation; cerebellum; gamma rhythms
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Other): healthy subjects will receive either sham or active cerebellar stimulation
  Interventions: Other: active cerebellar stimulation; Other: sham cerebellar stimulation
- Dystonia (Other): dystonic patients will receive either sham or active cerebellar stimulation
  Interventions: Other: active cerebellar stimulation; Other: sham cerebellar stimulation

INTERVENTIONS:
Other: active cerebellar stimulation
Other: sham cerebellar stimulation

SUMMARY:
Dystonia, a disabling disease with uncontrolled movement disorders was considered to be a manifestation of basal ganglia dysfunction, yet there is accumulating evidence from animal and human experiments that the cerebellum plays a prominent role in the pathophysiology of dystonia. Our recent results suggest a deficient cerebellar sensory encoding in dystonia, resulting in a decoupling of the motor component from the afferent information flow resulting from changes in the environment. An overall loss of gabaergic-mediated inhibition is at the forefront in dynamic changes in neural circuitry described in dystonia. In the mature brain gabaergic control the generation of temporal synchronies and oscillations in the glutamatergic neurons. Taken these all together with the results of a pilot experiment, the investigators hypothesize that deficient synchronies in the fast gamma range are one of the key mechanisms leading to abnormal communication inside the cerebello-cortical network in dystonia. The investigators aim first to demonstrate it by means of MEG (Magneto encepholography) recordings allowing to reconstruct the spatio-temporal dynamics of gamma oscillations in the nodes of the cerebello-cortical network. The investigators then aim to re-establish (if lost) or boost (if decreased) the defective synchronies by applying to the cerebellum at high gamma frequency a non invasive transcranial alternative current stimulation.

ELIGIBILITY:
Inclusion Criteria:

* primary upper limb dystonia
* normal physical and neurological examination except for dystonia
* no treatment with botulinum toxin during the three months preceding the study

Exclusion Criteria:

* Writing tremor
* current neurological or psychiatric illness other than dystonia
* uncontrollable medical problems not related to dystonia
* pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
change in gamma oscillations power in the cerebellum during a sensorimotor adaptation task | measures will be done at each of 3 visits: visit1, visit2 at expected average 7 days after visit1 and visit3 at expected average 14 days after visit1
  MEG recording will be performed using a whole-head 306-channels MEG system (Elekta Neuromag® TriuxTM System) comprising 204 planar gradiometers and 102 magnetometers regularly distributed at 102 locations over the scalp. MEG data will be coregistered with the structural MRI of each subject using BrainStorm (http://neuroimage.usc.edu/brainstorm).
  The localization of the source will be constrained with the individual anatomy obtained with MRI.

SECONDARY OUTCOMES:
synchrony in the gamma band between the cerebellum and the sensorimotor cortex | measures will be done at each of 3 visits: visit1, visit2 at expected average 7 days after visit1 and visit3 at expected average 14 days after visit1
  We will also conduct a functional connectivity analysis to assess the neuronal interactions between the cerebellum and the thalamus, the thalamus and the motor cortex by quantifying correlations between power envelopes. We will compute Pearson's linear correlation between the power envelopes from two different locations (between couples of magnetometers and couples of nodes at the source level).

OTHER OUTCOMES:
behavioral performances at a sensorimotor adaptation task | measures will be done at each of 3 visits: visit1, visit2 at expected average 7 days after visit1 and visit3 at expected average 14 days after visit1
  Subjects will have to reach six different targets positioned on a half-circle and appearing in a predictable order on a computer screen by moving a amagnetic joystick with their right hand. During the direct condition, there will be a direct coupling between the joystick and the cursor position. During the indirect conditions, 4 different rotations between the joystick and the cursor positions will be introduced. During one session the shifts will be 10°, 30°, -20°, -40° and in the other session -10°, -30°, 20°, 40° in order to reduce possible skill transfer from the baseline session to the stimulation session. Indirect and direct trials will be randomized to avoid habituation and learning within a session. There will be 2 blocks of 160 trials. In each block, there will be 20 trials for each rotation and 80 trials of the direct condition

CONTACTS AND LOCATIONS:
Overall Officials: sabine meunier, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- ICM GH Pitié Salpetrière, Paris, France